CLINICAL TRIAL: NCT02813434
Title: Cerebral Amyloid Imaging Using Florbetapir (18F-AV-45) for the Etiological Diagnosis of Poststroke Cognitive Impairment and Dementia
Brief Title: Cerebral Amyloid Imaging Using Florbetapir (AV-45)
Acronym: IDEA3
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2013_843_0011
Record Dates: First submitted 2016-06-20; First posted 2016-06-27 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Dementia; Cognition Disorders
Keywords: Cerebral amyloid imaging; Florbetapir; 18F-AV-45; poststroke
MeSH Terms: conditions — Dementia; Cognition Disorders | interventions — florbetapir

ARMS (1):
- Florbetapir (Experimental)
  Interventions: Biological: florbetapir

INTERVENTIONS:
Biological: florbetapir — 18F-AV-45 or 18F-Florbetapir

SUMMARY:
This study is aimed at examining the interest of amyloid radiotracer Florbetapir (18F-AV-45) for the etiological diagnosis of poststroke cognitive impairment and dementia

DETAILED DESCRIPTION:
This study is aimed at examining the interest of amyloid radiotracer Florbetapir (18F-AV-45) for the etiological diagnosis of poststroke cognitive impairment and dementia. This study stems from two converging objectives: (1) the need to refine characteristics of vascular cognitive impairment (VCI) and dementia (VD) in order to propose diagnosis criteria of VCI and of mixed dementia and to improve diagnosis criteria of VD and (2) the need to improve the etiological diagnosis of poststroke cognitive impairment and dementia. It will take advantage from the ongoing GRECOG-VASC study (which determines the cognitive status 6 months poststroke in consecutive patients according to a standardized international battery) coordinated by the Amiens University Hospital center, the opportunity to perform amyloid imaging in vivo using Positron Emission Tomography (PET) and Florbetapir (a production site is located in the city of Amiens) and the collaboration between neurology and imaging departments of Amiens University hospital.

ELIGIBILITY:
Inclusion Criteria:

1. patients suffering of parenchymal stroke visualized by imaging (MRI),
2. patients suffering from cognitive impairment on the 6 months assessment (including GRECogVASC patients),
3. age between 40 and 80 years,
4. French-speaking,
5. reliable informant,
6. agreeing to participate in the study,
7. affiliation to a social security system,

Exclusion Criteria:

1. women of childbearing potential (defined as pre-menopausal, less than 2 years postmenopausal, or not surgically sterile), or who are breast-feeding
2. history of relevant severe drug allergy or hypersensitivity,
3. patient receiving any investigational medications at least in the 30 last days,
4. stroke affecting the cerebellum,
5. mental retardation,
6. illiteracy,
7. dementia diagnosed before stroke,
8. history of schizophrenia or psychiatric illness requiring a stay for > 2 days in a psychiatry unit,
9. persons placed under judicial protection,
10. comorbidities affecting cognition (respiratory, renal, liver, heart failure),
11. persistent disturbance of consciousness defined by a score to item 1a of the National Institute of Health Stroke Scale (NIHSS) ≤ 1,
12. contraindication to MRI.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
presence of positive amyloid retention | 12 months
  determine the frequency of abnormal amyloid retention using PET with 18F-AV-45 on patients with poststroke cognitive impairment

SECONDARY OUTCOMES:
Final diagnosis | 12 months
  cognitive impairment or dementia

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GODEFROY, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

REFERENCES:
- [Derived] Godefroy O, Trinchard N, Marchal E, Lamy C, Canaple S, Meyer ME, Roussel M, Wollenweber FA; IDEA3 Study Group. Do Amyloid Cerebral Deposits Influence the Long-Term Poststroke Cognitive Outcome?: The IDEA3 Study. Stroke. 2025 Jan;56(1):74-83. doi: 10.1161/STROKEAHA.124.049147. Epub 2024 Dec 9. PMID 39648884